CLINICAL TRIAL: NCT06548958
Title: A Single-Arm, Prospective Clinical Study of Total Body Irradiation Combined With Busulfan and Melphalan (TBI+BUMEL) as a Conditioning Regimen for Second Hematopoietic Stem Cell Transplantation in Patients With Malignant Hematologic Diseases
Brief Title: A Single-Arm, Prospective Study of TBI+BUMEL as Conditioning for SCT2 in Patients With Malignant Hematologic Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOOCHOW-WXJ-2024-248
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-07

CONDITIONS: Malignant Hematological Diseases
Keywords: Second Allogeneic Hematopoietic Stem Cell Transplantation; Malignant Hematological Diseases; Total Body Irradiation; Melphalan; Conditioning Regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 40 patients with malignant hematological diseases who undergo SCT2 (Experimental): patients undergo SCT2 using TBI + BUMEL as a conditioning regimen
  Interventions: Procedure: Second Stem Cell Transplantation (SCT2)

INTERVENTIONS:
Procedure: Second Stem Cell Transplantation (SCT2) — 1. Conditioning Regimen Day -7: Semustine (Me-CCNU) 250mg/m², orally; Day -6: Total Body Irradiation (TBI) 4Gy; Day -5 to Day -4: Busulfan (Bu) 3.2mg/kg/day, administered in four divided doses, IV infusion; Day -3 to Day -2: Melphalan (Mel) 50mg/m²/day, IV infusion;
  2. Donor Stem Cell Infusion (Second Hematopoietic Stem Cell Transplantation) Day 0: Intravenous infusion of donor hematopoietic stem cells (MNC ≥ 8×10⁸/kg, CD34+ cells ≥ 4×10⁶/kg).

SUMMARY:
Each year, over 20,000 patients in China undergo hematopoietic stem cell transplantation (HSCT). Unfortunately, the prognosis in patients with disease relapse or graft failure is often inferior. A second allogeneic hematopoietic stem cell transplantation (SCT2) has emerged as a vital salvage therapy option. Despite varying prognoses, most patients undergoing SCT2 have a five-year overall survival (OS) rate of less than 30%. The primary challenges of SCT2 include treatment strategy, immune regulation, complication management, and transplantation technique improvements. By optimizing these key aspects, SCT2 can effectively address issues that arose after the first transplant, reduce complications, and provide more effective treatment for patients.

Clinical practice indicates that SCT2 is crucial in treating various hematologic diseases. For patients who failed the first transplant (SCT1), SCT2 can more effectively treat the primary disease, provide timely hematopoietic engraftment, extend survival time, and improve the quality of life. Additionally, the successful application of SCT2 provides clinicians with more treatment options and hope. Currently, the modified BU/CY conditioning regimen, which consists of busulfan (BU) and cyclophosphamide (CY), is commonly used in SCT1 in China. However, for patients who relapse after SCT1, these drugs may become ineffective, and the physical condition often worsens, with a higher likelihood of infections and organ dysfunction. Therefore, finding new conditioning regimens is crucial.

Studies have shown that a melphalan (MEL)-based conditioning regimen may have better outcomes for patients with acute myeloid leukemia (AML) compared to a Cy-based regimen. The Conditioning regimen that includes total body irradiation (TBI) has also been considered effective for patients with acute leukemia. Thus, low-dose TBI combined with a BU + MEL regimen could be a promising conditioning regimen for SCT2. In the investigators' preliminary studies, three patients who underwent SCT2 with this regimen successfully achieved engraftment and were discharged.

Based on this, the investigators plan to conduct a clinical study to observe the effects of the TBI+BUMEL regimen combined with SCT2 on the engraftment rate, disease relapse rate, GVHD incidence, and survival rate in patients with malignant hematologic diseases who relapsed after SCT1.

DETAILED DESCRIPTION:
The primary challenges of SCT2 include:

1. treatment strategy: eliminating residual tumor cells and addressing graft failure;
2. immune regulation: adjusting the immune system to ensure successful engraftment of new stem cells;
3. complication management: due to the poor physical condition of patients after the first transplant (SCT1), the risk of complications after SCT2 is high. This necessitates special attention to the prevention and management of post-transplant complications;
4. transplantation technique improvements: more rigorous donor screening, HLA typing, monitoring, and supportive treatment during the transplant procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Gender is not limited, patients between 14 to 70 years old (including critical value);
2. Malignant hematological diseases (acute/chronic myeloid leukemia, acute lymphoblastic leukemia, myelodysplastic syndrome, malignant lymphoma, etc.) diagnosed by bone marrow aspiration or biopsy according to the WHO diagnostic criteria, after the first hematopoietic stem cell transplantation, due to various reasons (including but not limited to disease relapse or graft failure) have indications for a second hematopoietic stem cell transplantation;
3. The indexes of cardiac function, liver and kidney function were within the following limits: (1) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3× Upper limit of normal (ULN); (2)Total bilirubin ≤ 3×ULN; (3) Serum creatinine ≤ 2×ULN or creatinine clearance ≥ 40mL/min; (4) Left ventricular ejection fraction (LVEF) as measured by echocardiography or multi-gated acquisition (MUGA) scan is within the normal range (> 50%);
4. Having a suitable allogeneic hematopoietic stem cell donor;
5. Expected survival ≥3 months;
6. Karnofsky (KPS) score ≥60%, Eastern Tumor Cooperative group (ECOG) status ≤ 2;
7. Patient fully understood the nature of the study, and voluntarily participates and signs informed consent.

Exclusion Criteria:

1. Patients had serious adverse reactions to investigational drugs such as allergies;
2. Patients with a history of immunodeficiency, or other acquired or congenital diseases, immunodeficiency diseases, and a history of organ transplantation;
3. Patients with hypertension, ventricular arrhythmia requiring clinical intervention, acute coronary syndrome, congestive heart failure, stroke, or other grade III or higher cardiovascular events within 6 months;
4. Received Class II or higher surgery within 4 weeks prior to enrollment;
5. Patients with active viral infections;
6. Pregnant or lactating patients;
7. The patient is currently participating in another clinical studies;
8. Patients deemed unsuitable for inclusion by other investigators.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The cumulative incidence of neutrophil engraftment and platelet engraftment | on day 28±7 following SCT2
  Neutrophil and platelet engraftment is defined as the first occurrence of 3 consecutive days with an absolute neutrophil count of at least 0.5×109/L and a platelet count of over 20×109/L for 7 consecutive days without transfusion support.
The time to reconstitution of hematopoiesis | on day 28±7 following SCT2
  Recovery of hemopoietic function after treatment
The cumulative incidence of transplant-related mortality (TRM) | within 100 days following SCT2
  Transplant-related mortality was defined as mortality due to any cause other than disease progression within 100 days of transplantation.

SECONDARY OUTCOMES:
The cumulative incidence and grade of graft-versus-host disease (GVHD) | within 1 year following SCT2
  Graft-versus-host disease (GvHD) is a medical complication following the receipt of transplanted tissue from a genetically different person.
The cumulative incidence of relapse | within 1 year following SCT2
  We defined relapse as any clinical evidence of progression or recurrence of original diseases.
Overall survival rate | within 1 year following SCT2
  We estimated OS from the time of transplant until the date of death of any cause or last follow-up for patients still alive.
The cumulative incidence of adverse events | within 1 year following SCT2
  Following extraction of the tumor, a blood vessel burst causing increased blood loss during the procedure, an adverse event the surgeon did not expect.

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, Prof., Principal Investigator — The First Affiliated Hospital of Soochow University; Xiaojin Wu, Prof., Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- Hematology Department, The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China